CLINICAL TRIAL: NCT01810393
Title: An Open-Label, Randomized, Multicenter Phase III Study in Patients With HER2-Positive Metastatic Breast Cancer Responding to First Line Treatment With Intravenous Trastuzumab for at Least 3 Years and Investigating Patient Preference for Subcutaneous Trastuzumab
Brief Title: A Study to Assess Preference for Subcutaneous Trastuzumab Treatment in Participants With Human Epidermal Growth Factor Receptor (HER)2-Positive Metastatic Breast Cancer Responding to First-Line Intravenous Trastuzumab for at Least 3 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ML28589; 2012-003442-32 (EudraCT Number)
Record Dates: First submitted 2013-03-11; First posted 2013-03-13 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

ARMS (2):
- Trastuzumab IV Then Trastuzumab SC (Experimental): Participants will receive treatment with Trastuzumab IV for the first 3 cycles (cycle length = 21 days) followed by Trastuzumab SC for the next 3 cycles. Participants will continue receiving treatment with trastuzumab SC for another 12 cycles (if SC treatment is well tolerated, otherwise participants will continue IV treatment) for a total of 18 cycles of treatment during the study.
  Interventions: Drug: Trastuzumab
- Trastuzumab SC Then Trastuzumab IV (Experimental): Participants will receive treatment with Trastuzumab SC for the first 3 cycles (cycle length = 21 days) followed by Trastuzumab IV for the next 3 cycles. Participants will continue receiving treatment with trastuzumab SC for another 12 cycles (if SC treatment is well tolerated, otherwise participants will continue IV treatment) for a total of 18 cycles of treatment during the study.
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab — Trastuzumab will be administered at a dose of 6 milligrams per kilogram (mg/kg) IV or 600 milligrams per 5 milliliter (mg/5mL) SC in 21-day cycles as per schedule described in respective arm.
  Other Names: Herceptin

SUMMARY:
This open-label, randomized, multicenter study will evaluate participant preference for subcutaneous (SC) versus intravenous (IV) trastuzumab (Herceptin) in participants with HER2-positive metastatic breast cancer responding to first-line treatment with IV trastuzumab for at least 3 years. Participants will be randomized to receive either 3 cycles (cycle length = 21 days) of trastuzumab SC followed by 3 cycles of trastuzumab IV or 3 cycles of trastuzumab IV followed by 3 cycles of trastuzumab SC. All participants will receive trastuzumab SC for Cycles 7 to 18. Anticipated time on study treatment is 1 year or until disease progression or inacceptable toxicity occurs, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed HER2-positive metastatic breast cancer
* On treatment with first-line trastuzumab IV and free of disease progression for at least 3 years
* Left ventricular ejection fraction (LVEF) of greater than or equal to (>/=) 50 percent (%)
* Hormonal therapy will be allowed
* Prior use of anti-HER2 therapy will be allowed

Exclusion Criteria:

* History of other malignancy, except for curatively treated carcinoma in situ of the cervix or basal cell carcinoma and participants with other curatively treated malignancies who have been disease-free for at least 5 years; participants with previous ductal carcinoma in situ of the breast are also eligible
* Participants with severe dyspnea at rest or requiring supplementary oxygen therapy
* Serious cardiac illness or medical conditions that would preclude the use of trastuzumab
* Hepatitis B, hepatitis C or human immunodeficiency virus infection
* Pregnant or lactating women
* Concurrent enrollment in an other clinical trial using an investigational anti-cancer treatment, including hormonal therapy, biphosphonate therapy and immunotherapy, within 28 days prior to the first dose of study treatment
* Known hypersensitivity to trastuzumab, murine proteins, to any of the excipients of Herceptin including hyaluronidase or the adhesive of the subcutaneous device, or a history of severe allergic or immunological reactions, for example, difficult to control asthma
* Central nervous system metastases, unless they have been treated and have been stable for at least 3 years
* Inadequate organ function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2013-06-11 (Actual); Primary Completion 2019-07-17 (Actual); Study Completion 2019-07-17 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Preference for Either SC or IV Route of Administration According to Participant Preference Questionnaire (PPQ) Score | Baseline up to 6 cycles (cycle length = 21 days)

SECONDARY OUTCOMES:
Percentage of Participants With Adverse Events | approximately 4 years
Percentage of Health Care Professionals With Preference for Either SC or IV Administration According to Health Care Professional Questionnaire (HCPQ) Score | Baseline up to 6 cycles (cycle length = 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (61):
- France (61):
  - Clinique Du Docteur Calabet; Cromg, Agen
  - Clinique De L Europe; Radiotherapie Chimiotherapie, Amiens
  - ICO Paul Papin; Oncologie Medicale., Angers
  - HOP Prive Arras Les Bonnettes; Chimiotherapie, Arras
  - Institut Sainte-Catherine; Oncologie, Avignon
  - Centre Hospitalier de La Cote Basque; Oncologie, Bayonne
  - HOPITAL JEAN MINJOZ; Oncologie, Besançon
  - Institut Bergonie, Bordeaux
  - Centre Hospitalier Fleyriat; Oncologie/Hematologie, Bourg-en-Bresse
  - Hopital Morvan, Brest
  - Clinique Pasteur Lanroze; Chimiotherapie Radiotherapie, Brest
  - Centre Francois Baclesse; Oncologie, Caen
  - Centre Jean Perrin; Oncologie, Clermont-Ferrand
  - Pole Sante Republique;Oncologie Hematologie, Clermont-Ferrand
  - Chi De Creteil; Radiotherapie Oncologie, Créteil
  - Centre Leonard De Vinci;Chimiotherapie, Dechy
  - Centre Georges Francois Leclerc; Oncologie 3, Dijon
  - CHD Les Oudairies, La Roche-sur-Yon
  - Ch Louis Pasteur; Oncologie, Le Coudray
  - Clinique Victor Hugo; Radiotherapie, Le Mans
  - Polyclinique Du Bois; Oncologie, Lille
  - Centre Oscar Lambret; Unite de Recherche Clinique, Lille
  - Ch Bretagne Sud Site Scorff; Oncologie Medicale, Lorient
  - Centre Leon Berard, Lyon
  - Clinique De La Sauvegarde; Chimiotherapie, Lyon
  - Hopital Prive Jean Mermoz, Lyon
  - Institut Paoli Calmettes; Oncologie Medicale, Marseille
  - Hopital de Mercy ;ONCOLOGIE MEDICALE, Melz-sur-Seine
  - Hopital Belle Isle; Oncologie Hematologie, Metz
  - Clinique Clementville; Hopital De Jour, Montpellier
  - Polyclinique Gentilly; CHIMIOTHERAPIE AMBULATOIRE, Nancy
  - Centre Catherine de Sienne; Chimiotherapie, Nantes
  - Centre Antoine Lacassagne, Nice
  - Institut de cancerologie du Gard, Nîmes
  - HOPITAL DE LA SOURCE; Service de Cardiologie, Point Jaune, Orléans
  - APHP - Hopital de la Pitie Salpetriere, Paris
  - Groupe Hospitalier Diaconesses, Paris
  - Institut Curie; Oncologie Medicale, Paris
  - Hopital Saint Louis; Oncologie Medicale, Paris
  - HOPITAL TENON; Cancerologie Medicale, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - CH d'Annecy, Pringy
  - Chi De Cornouaille; Oncologie Hospitalisation, Quimper
  - Institut Jean Godinot; Oncologie Medicale, Reims
  - Institut du Cancer Coulancy Reims, Reims
  - Centre Eugene Marquis; Bureau D Etudes Cliniques, Rennes
  - Centre Henri Becquerel; Oncologie Medicale, Rouen
  - Chp Saint Gregoire; Cancerologie Radiotherapie, Saint-Grégoire
  - Centre Rene Gauducheau, Saint-Herblain
  - Polyclinique de la Cote Basque Sud; Oncologie, Saint-Jean-de-Luz
  - CMCO De La Cote D Opale; Auberge De Jour, Saint-Martin-Boulogne
  - Clinique Mutualiste L Estuaire, Saint-Nazaire
  - Institut de Cancérologie de Loire, Saint-Priest-en-Jarez
  - CH de Saint Quentin, Saint-Quentin
  - Hopital Prive Nord Parisien; Soins De Suite - Oncologie, Sarcelles
  - Clinique Ste Anne, Strasbourg
  - Centre Paul Strauss; Oncologie Medicale, Strasbourg
  - Hopital de Hautepierre, Strasbourg
  - Hôpital Rangueil - CHU de Toulouse, Toulouse
  - Clinique Pasteur; Oncologie Medicale, Toulouse

REFERENCES:
- [Derived] Pivot X, Spano JP, Espie M, Cottu P, Jouannaud C, Pottier V, Moreau L, Extra JM, Lortholary A, Rivera P, Spaeth D, Attar-Rabia H, Benkanoun C, Dima-Martinez L, Esposito N, Gligorov J. Patients' preference of trastuzumab administration (subcutaneous versus intravenous) in HER2-positive metastatic breast cancer: Results of the randomised MetaspHer study. Eur J Cancer. 2017 Sep;82:230-236. doi: 10.1016/j.ejca.2017.05.009. Epub 2017 Jun 23. PMID 28648618